CLINICAL TRIAL: NCT02667223
Title: A Phase 1, Open Label, Randomized, Single Dose, Dose Escalation Study To Assess The Subcutaneous Pharmacokinetics And Pharmacodynamics Of Bococizumab (pf 04950615) Alone And In Co Mixture With Recombinant Human Hyaluronidase (rhuph20, Pf 06744547) In Healthy And Hypercholesterolemic Adult Subjects
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Bococizumab Alone and When Combined With Recombinant Human Hyaluronidase
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early on July 8, 2016 due to business priorities regarding study execution.
Sponsor: Pfizer (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: B1481051; 2015-003568-36 (EudraCT Number)
Record Dates: First submitted 2016-01-06; First posted 2016-01-28 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Healthy; Hypercholesterolemia
Keywords: pharmacokinetics; pharmacodynamics; RN316; recombinant human hyaluronidase
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: bococizumab 150 mg + rHuPH20 (Experimental): bococizumab 150 mg co-mixed with rHuPH20 and administered subcutaneously to healthy volunteers
  Interventions: Biological: Cohort 1: bococizumab 150 mg + rHuPH20
- Cohort 2: bococizumab 300 mg (Active Comparator): bococizumab 300 mg administered subcutaneously to healthy volunteers
  Interventions: Biological: Cohort 2: bococizumab 300 mg
- Cohort 3: bococizumab 300 mg + rHuPH20 (Experimental): bococizumab 300 mg co-mixed with rHuPH20 and administered subcutaneously to healthy volunteers
  Interventions: Biological: Cohort 3: bococizumab 300 mg + rHuPH20
- Cohort 5: bococizumab 450 mg + rHUPH20 (Experimental): bococizumab 450 mg co-mixed with rHuPH20 and administered subcutaneously to healthy volunteers
  Interventions: Biological: Cohort 5: bococizumab 450 mg + rHuPH20
- Cohort 4: bococizumab 300 mg + rHuPH20 (Experimental): bococizumab 300 mg co-mixed with rHuPH20 and administered subcutaneously to subjects with hypercholesterolemia receiving a statin
  Interventions: Biological: Cohort 4: bococizumab 300 mg + rHuPH20

INTERVENTIONS:
Biological: Cohort 1: bococizumab 150 mg + rHuPH20 — bococizumab 150 mg + rHuPH20 administered SC to healthy volunteers
  Arms: Cohort 1: bococizumab 150 mg + rHuPH20
Biological: Cohort 2: bococizumab 300 mg — bococizumab 300 mg administered SC to healthy volunteers
  Arms: Cohort 2: bococizumab 300 mg
Biological: Cohort 3: bococizumab 300 mg + rHuPH20 — bococizumab 300 mg + rHuPH20 administered SC to healthy volunteers
  Arms: Cohort 3: bococizumab 300 mg + rHuPH20
Biological: Cohort 5: bococizumab 450 mg + rHuPH20 — bococizumab 450 mg + rHuPH20 administered SC to healthy volunteers
  Arms: Cohort 5: bococizumab 450 mg + rHUPH20
Biological: Cohort 4: bococizumab 300 mg + rHuPH20 — bococizumab 300 mg + rHuPH20 administered SC to subjects with hypercholesterolemia receiving a statin
  Arms: Cohort 4: bococizumab 300 mg + rHuPH20

SUMMARY:
This is a Phase 1, open-label, single-dose, randomized, dose escalation study in healthy and hypercholesterolemic subjects. Each subject will receive 1 of 5 treatments as a single subcutaneous injection. Subjects will remain confined at the research clinic for approximately 2 days. After discharge, subjects will return to the research clinic 15 times during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and hypercholesterolemic subjects between the ages of 18 and 65 years.
* Healthy subjects must have fasting LDL-C >/= 70 to </= 190 mg/dL at two qualifying visits.
* Hypercholesterolemic subjects must be on a stable daily dose of statin for at least 45 days before dosing and fasting LDL-C must be >/= 70 mg/dL.

Exclusion Criteria:

* Use of prescription or non-prescription drugs within 7 days or 5 half-lives (whichever) is longer prior to the first dose of study medication. For hypercholesterolemic subjects the use of statin class medication is allowed.
* Prior exposure to bococizumab (also known as PF-04950615 or RN316) or other investigational PCSK9 inhibitors.
* Treatment with monoclonal antibodies within 6 months or 5 half-lives (whichever is longer) before dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
AUCinf of bococizumab | Day 1 - Day 85
  Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞), if data permits (otherwise AUClast will be used).
Cmax of bococizumab | Day 1 - Day 85
  Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Tmax | Day 1 - Day 85
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
CL/F | Day 1 - Day 85
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance is influenced by the fraction of the dose absorbed. Clearance is estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Vz/F | Day 1 - Day 85
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after dose (Vz/F) is influenced by the fraction absorbed.
t1/2 | Day 1 - Day 85
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
LDL-C at Week 4 | Baseline to Week 4
  Absolute value, and absolute change and % change in LDL cholesterol at Week 4 following bococizumab administration alone and when co-mixed with rHuPH20.
MaxELDL-C | Baseline up to Day 85
  Maximum LDL-C lowering calculated using absolute LDL-C values
Tmax, LDL-C | Baseline up to Day 85
  Time to MaxELDL-C calculated using absolute LDL-C values
AUEC85 | Baseline up to Day 85
  Area under the LDL-C concentration-time curve calculated using absolute LDL-C values
AEs | Baseline up to Day 85
  Incidence, severity, and causal relationship of treatment-emergent adverse events (TEAEs)
Laboratory tests | Baseline up to Day 85
  Incidence of abnormal and clinically relevant safety laboratory tests including clinical chemistry and hematology
Vital signs | Baseline up to Day 85
  Incidence of abnormal and clinically relevant vital signs
AUClast of bococizumab | Day 1 - Day 85
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
ADA | Day 1 - Day 85
  Incidence and titer of Anti-Drug Antibodies (ADA) following administration of bococizumab alone and when co-mixed with rHuPH20.
nAb | Day 1- Day 85
  Incidence and titer of neutralizing antibodies (nAb), if applicable, following administration of bococizumab alone and when co-mixed with rHuPH20.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Bass A, Plotka A, Mridha K, Sattler C, Kim AM, Plowchalk DR. Pharmacokinetics, pharmacodynamics, and safety of bococizumab, a monoclonal antibody against proprotein convertase subtilisin/kexin type 9, in healthy subjects when administered in co-mixture with recombinant human hyaluronidase: A phase 1 randomized trial. Health Sci Rep. 2018 Jul 18;1(9):e61. doi: 10.1002/hsr2.61. eCollection 2018 Sep. PMID 30623096
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481051&StudyName=A%20Phase%201%2C%20Open%20Label%2C%20Randomized%2C%20Single%20Dose%2C%20Dose%20Escalation%20Study%20To%20Assess%20The%20Subcutaneous%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Bococizumab%20%28pf%2004950615%29%20Alone%20And%20In%20Co%20Mixture%20With%20Recombinant%20Human%20Hyaluronidase%20%28rhuph20%2C%20Pf%2006744547%29%20In%20Healthy%20And%20Hypercholesterolemic%20Adult%20Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481051&StudyName=A+Phase+1%2C+Open+Label%2C+Randomized%2C+Single+Dose%2C+Dose+Escalation+Study+To+Assess+The+Subcutaneous+Pharmacokinetics+And+Pharmacodynamics+Of+Bococizumab+%28pf+04950615%29+Alone+And+In+Co+Mixture+With+Recombinant+Human+Hyaluronidase+%28rhuph20%2C+Pf+06744547%29+In+Healthy+And+Hypercholesterolemic+Adult+Subjects